CLINICAL TRIAL: NCT01753908
Title: A Pilot Study of Broccoli Sprout Extract in Patients With Breast Cancer
Brief Title: Broccoli Sprout Extract in Treating Patients With Breast Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: I 211911; NCI-2012-01770 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 211911 (Other: Roswell Park Cancer Institute); K07CA148888 (NIH); P30CA016056 (NIH)
Record Dates: First submitted 2012-12-10; First posted 2012-12-20 (Estimated); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Ductal Breast Carcinoma; Ductal Breast Carcinoma In Situ; Estrogen Receptor Negative; Estrogen Receptor Positive; Invasive Breast Carcinoma; Lobular Breast Carcinoma; Postmenopausal; Stage IA Breast Cancer; Stage IB Breast Cancer; Stage IIA Breast Cancer; Stage IIB Breast Cancer
MeSH Terms: conditions — Carcinoma, Ductal, Breast; Carcinoma, Intraductal, Noninfiltrating; Carcinoma, Lobular; Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (broccoli sprout extract) (Experimental): Patients receive broccoli sprout extract PO QD on days 1-14 immediately prior to surgery.
  Interventions: Drug: Broccoli Sprout Extract; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study
- Arm II (placebo) (Placebo Comparator): Patients receive placebo PO QD on days 1-14 immediately prior to surgery.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Other: Placebo

INTERVENTIONS:
Drug: Broccoli Sprout Extract — Given PO
  Arms: Arm I (broccoli sprout extract)
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Urinary ITCs and metabolites measured
Other: Placebo — Given PO
  Other Names: placebo therapy; PLCB; sham therapy
  Arms: Arm II (placebo)

SUMMARY:
This randomized pilot trial studies broccoli sprout extract in treating patients with breast cancer. Broccoli sprout extract contains ingredients that may prevent or slow the growth of certain cancers. Studying samples of tissue from patients receiving broccoli sprout extract may help determine if it can enter breast tumor cells and how it affects certain biomarkers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether isothiocyanate-rich broccoli sprout extract (ITC-BSE) modifies biomarkers in breast tumor cells.

II. To determine whether the intervention alters proliferative and apoptotic markers (Ki-67 and cleaved caspase-3).

III. To determine whether the intervention down-regulates the expression of estrogen receptor (ER) including both ERalpha and ERbeta.

IV. To determine whether the intervention induces NAD(P)H dehydrogenase (quinone) 1 (NQO1) expression.

SECONDARY OBJECTIVES:

I. To determine tolerability of ITC-BSE and compliance in breast cancer patients.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive broccoli sprout extract orally (PO) once daily (QD) on days 1-14 immediately prior to surgery.

ARM II: Patients receive placebo PO QD on days 1-14 immediately prior to surgery.

After completion of study treatment, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal (no menstrual cycle in the past 12 months)
* Diagnosed with incident, primary, invasive, ductal or lobular, or other epithelial malignancy, clinical stage I or II, ER positive or negative breast cancer, or ductal carcinoma in situ (DCIS)
* No neoadjuvant endocrine therapy or chemotherapy within 12 months
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of =< 2
* Willing to avoid cruciferous vegetable intake during the study period (2 weeks)
* Demonstrate the ability to swallow and retain oral medication
* Subject or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Prior invasive breast cancer, prior mastectomy or breast radiation within 12 months
* Current or recent use of reproductive hormone therapy, tamoxifen, aromatase inhibitor or other estrogen inhibitors within the last 90 days, which may affect biomarkers
* Intolerance to broccoli/ITC-BSE taste
* Current ingestion of broccoli sprout extract, which may confound study results
* Current or recent treatment for any malignancy within the last one year, which may affect biomarkers
* History of Crohn's disease, celiac sprue or other malabsorption syndrome which may interfere with digestion and absorption of broccoli sprout extract
* Current diagnosis of Gastroesophageal Reflux Disease (GERD) with grade >3

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-05-21 (Actual); Primary Completion 2018-07-23 (Actual); Study Completion 2018-08-23 (Actual)

PRIMARY OUTCOMES:
Changes in apoptosis (cleaved caspase 3) | Baseline to up to 14 days
  Appropriate transformation (such log transformation) will be used to achieve normality of the data. Results will be given as the back-transformed geometric means and 95% confidence intervals in order to preserve the units of measurement. Change in immunohistochemistry measures will be calculated for each individual and compared between treatment and placebo groups by use of independent samples t-test. If the normality could not be reached by transformation, Wilcoxon rank-sum test will be used, which considers both the direction and the magnitude of changes.
Changes in cell proliferation (Ki-67) | Baseline to up to 14 days
  Appropriate transformation (such log transformation) will be used to achieve normality of the data. Results will be given as the back-transformed geometric means and 95% confidence intervals in order to preserve the units of measurement. Change in immunohistochemistry measures will be calculated for each individual and compared between treatment and placebo groups by use of independent samples t-test. If the normality could not be reached by transformation, Wilcoxon rank-sum test will be used, which considers both the direction and the magnitude of changes.
Changes in estrogen receptor expression (ER alpha and ER beta) | Baseline to up to 14 days
  Appropriate transformation (such log transformation) will be used to achieve normality of the data. Results will be given as the back-transformed geometric means and 95% confidence intervals in order to preserve the units of measurement. Change in immunohistochemistry measures will be calculated for each individual and compared between treatment and placebo groups by use of independent samples t-test. If the normality could not be reached by transformation, Wilcoxon rank-sum test will be used, which considers both the direction and the magnitude of changes.
Changes in NQO1 expression | Baseline to up to 14 days
  Appropriate transformation (such log transformation) will be used to achieve normality of the data. Results will be given as the back-transformed geometric means and 95% confidence intervals in order to preserve the units of measurement. Change in immunohistochemistry measures will be calculated for each individual and compared between treatment and placebo groups by use of independent samples t-test. If the normality could not be reached by transformation, Wilcoxon rank-sum test will be used, which considers both the direction and the magnitude of changes.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Young, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States